CLINICAL TRIAL: NCT06942507
Title: A Multicenter Study on the First-line Treatment of Waldenström's Macroglobulinemia With Zanubrutinib in Combination With Rituximab and Bendamustine
Brief Title: Zanubrutinib Combined With BR in the First-line Treatment of Waldenström's Macroglobulinemia
Acronym: BRZ-WM
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, Jian Li, Professor, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BRZ-WM
Record Dates: First submitted 2025-04-17; First posted 2025-04-24 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Waldenström's Macroglobulinemia (WM)
Keywords: Rituximab; Zanubrutinib; MYD88; Waldenström's Macroglobulinemia; Bendamustine
MeSH Terms: conditions — Waldenstrom Macroglobulinemia | interventions — zanubrutinib; Bendamustine Hydrochloride; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- BRZ (Experimental): participants recieve 4 to 6 cycles of the zanubrutinib-rituximab-bendamustine regimen
  Interventions: Drug: Zanubrutinib; Drug: Bendamustine + Rituximab

INTERVENTIONS:
Drug: Zanubrutinib — zanubrutinib 160mg po bid d1-28
Drug: Bendamustine + Rituximab — bendamustine 70-90mg/m2 ivgtt d1-2, rituximab 375mg/m2 ivgtt d1

SUMMARY:
Current retrospective studies have demonstrated that achieving deep remission following treatment for Waldenström's macroglobulinemia (WM) correlates with prolonged survival. While the bendamustine-rituximab (BR) regimen or single-agent zanubrutinib are currently recommended as first-line therapies, neither achieves optimal deep remission. Additionally, prolonged zanubrutinib monotherapy may lead to cumulative adverse effects. Therefore, this study aims to evaluate the efficacy and safety of the bendamustine-rituximab-zanubrutinib combination regimen as a first-line treatment option for MYD88-mutated WM patients.

ELIGIBILITY:
Inclusion Criteria:

1. Previously untreated symptomatic Waldenström macroglobulinemia (WM) meeting IWWM-7 diagnostic criteria:

   1. Presence of monoclonal IgM-type immunoglobulin in serum
   2. Bone marrow infiltration by plasmacytoid lymphocytes or bone marrow biopsy showing small lymphocytes/plasma cells/plasmacytoid lymphocytes (any quantity) in the intertrabecular space
   3. Exclusion of other non-Hodgkin lymphoma subtypes
   4. Typical immunophenotype: CD5-/CD10-/CD19⁺/CD20⁺/CD23-/CD79b⁺ /sIgM⁺/CD138- clonal B-cells. Variant phenotypes may show CD5/CD10/CD23 /CD38 positivity or coexistence of clonal B-cells and plasma cells.
2. MYD88 L265P mutation is detected in peripheral blood or bone marrow.
3. Serum monoclonal IgM ≥5 g/L.

Exclusion Criteria:

1. Co-morbidity of uncontrolled infection or autoimmune disease
2. Co-morbidity of other active malignancy
3. Co-morbidity of uncontrolled heart disease
4. Co-morbidity of severe digestive system disorders precluding oral medication
5. Seropositive for human immunodeficiency virus
6. Hepatitis B virus (HBV)-DNA > 1000 copies/mL
7. Seropositive for hepatitis C (except in the setting of a sustained virologic response)
8. Neutrophil <1×10E9/L, platelet < 75×10E9/L, alanine transaminase (ALT) or aspertate aminotransferase (AST) > 2.5 × upper limit of normal (ULN), total bilirubin > 1.5 × ULN，eGFR < 30 mL/min, or receiving renal replacement therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Estimated)
Dates: Start 2025-05-01 (Estimated); Primary Completion 2027-04-30 (Estimated); Study Completion 2029-04-30 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Achieving Complete Response (CR) at 4 to 6 Months After Treatment Initiation | 4 to 6 months after treatment initiation

SECONDARY OUTCOMES:
Number of Participants Achieving Very Good Partial Response (VGPR) at 4 to 6 Months After Treatment Initiation | 4 to 6 months after treatment initiation
Number of Participants Achieving Overall Response (OR) at 4 to 6 Months After Treatment Initiation | 4 to 6 months after treatment initiation
  CR + VGPR + partial response (PR)
Rate of Progression-Free Survival | 2 years
Time to next treatment | 2 years
Rate of Overall Survival | 2 years
Duration of response | 2 years

OTHER OUTCOMES:
Medical resource utilization | 4 to 6 months after treatment initiation

CONTACTS AND LOCATIONS:
Locations (1):
- Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No